CLINICAL TRIAL: NCT02588534
Title: An Open-label, Randomized, 2-period Crossover Bioequivalence Study Comparing a 50-mg Dose of Liquid Etanercept Administered to Healthy Subjects by Subcutaneous Injection in the Thigh Using an Auto-injector Device and Manual Injection
Brief Title: Open-label Study Using 50 Mg Liquid Etanercept Subcutaneous Injection in the Thigh to Compare an Auto-injector Device and a Manual Injection in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20040136
Record Dates: First submitted 2015-06-18; First posted 2015-10-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Healthy Men and Women
Keywords: etanercept, healthy subject,open-label, randomized, auto-injection, bioequivalence, pharmacokinetic
MeSH Terms: interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A-etanercept (ENBREL®) via auto-injector device (Active Comparator): Single dose of etanercept (ENBREL®) in a pre-filled syringe administered with an auto-injector device manufactured by Scandinavian Health Limited (SHL)
  Interventions: Device: etanercept (ENBREL®) via auto-injector device
- Treatment B-etanercept (ENBREL®) via Manual injection (Other): single dose of etanercept (ENBREL®) in a syringe given by manual injection (reference treatment)
  Interventions: Other: Etanercept (ENBREL®) via Manual injection

INTERVENTIONS:
Device: etanercept (ENBREL®) via auto-injector device — single 50 mg subcutaneous dose of liquid etanercept (ENBREL®) in a 1.0 ml pre-filled syringe administered via an auto-injector device manufactured by Scandinavian Health Limited (SHL)
  Arms: Treatment A-etanercept (ENBREL®) via auto-injector device
Other: Etanercept (ENBREL®) via Manual injection — single 50 mg subcutaneous dose of liquid etanercept (ENBREL®) in a 1.0 ml pre-filled syringe administered via manual injection (reference treatment) to compare to the auto-injection
  Arms: Treatment B-etanercept (ENBREL®) via Manual injection

SUMMARY:
A single-center, open-label, randomized study with a screening period of up to 21 days. Following that, eligible men and women will receive 50 mg of etanercept subcutaneously in the thigh to compare injection by auto-injection device to manual injection (each injection separated by 28 days)

DETAILED DESCRIPTION:
A single-center, open-label, 2-period, 2-sequence, 2-treatment, randomized, crossover study. After a screening period of up to 21 days before dosing, 36 eligible men and women will be assigned to receive a 50-mg subcutaneous (SC) dose of etanercept administered by each of 2 methods of injection (Treatment A: administration by auto-injector device; and Treatment B: administration by manual injection) on separate occasions in an order determined by a randomization list (randomized 1:1 to sequence). Treatment administrations will be separated by a minimum of 28 days (maximum of 36 days). Subjects will be required to remain resident during the 72-hours after dosing in each period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the age of 18 and 45 years, inclusive at the time of screening
* Body mass index (BMI) between 19 and 30 kg/m2, inclusive at the time of screening
* Absence of clinically significant physical examination findings as determined by the investigator and free of any clinically significant disease or condition that requires care by a physician that would interfere with the study evaluation or procedures
* 12-lead ECG (reporting ventricular rate and PR, QRS, QT and QTc intervals) within normal limits or clinically acceptable to the investigator
* Negative human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), and hepatitis C antibody (HepCAb) status at the time of screening
* Negative pregnancy test for all women at screening and the day before dosing
* Willing to reside in the research facility for 3 consecutive nights, on two occasions, and willing to return to research facility for scheduled follow-up visits
* Before any study specific procedures or administration of study medication, the subject must sign the Institutional Review Board (IRB)-approved informed consent form

Exclusion Criteria:

* Unstable medical condition, defined as having been hospitalized within 30 days, myocardial infarction within 6 months, major surgery within 6 months, or a seizure within 12 months of study day 1, or otherwise unstable in the judgment of the investigator (i.e., at risk of complications or adverse events unrelated to study participation)
* Clinically significant abnormality in chemistry, hematology, or urinalysis parameters performed at screening as determined by the investigator
* Current active infection, including chronic or localized infection or history of recurring infections with underlying condition that may predispose one to infection (e.g., diabetes)
* Known history of active tuberculosis
* Donated blood or blood products within 12 weeks before day -1, or a total of 1500 mL within 1 year before day -1
* Known hypersensitivity to etanercept or any excipients
* Use of any prescription or over-the-counter medication within 7 days before day -1 without the approval of the investigator (with the exception of vitamins, topical medications, contraceptive medications, or hormonal replacement therapy in postmenopausal women)
* Consumption of alcohol within 48 hours before dosing
* Known history of drug or alcohol abuse within 1 year of screening
* Positive urine screen for alcohol and/or potential drugs of abuse, at screening, and the day before dosing
* Smoked more than 10 cigarettes per day within the 12 months before day -1
* Women who are nursing or lactating
* Unwilling or unable to practice an adequate barrier method of contraception (e.g., condom, barrier method contraceptive with spermicide, IUD, etc.), as determined by the investigator, for the duration of the study
* Use of an investigational agent, drug, and/or device within 30 days of screening
* Any other condition that might reduce the chance of obtaining data (e.g., known poor compliance) required by the protocol or that might compromise the ability to give informed consent

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-08; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Ratio of the geometric mean of etanercept (ENBREL®) administered by auto-injector Scandinavian Health Limited-SHL) to etanercept administered by manual injection for the pharmacokinetic (PK) parameter of AUC(0-t) | 28 days following each treatment arm
  28 days after receiving treatment in Period 1, subjects return to the facility on an outpatient basis to receive the alternate treatment in Period 2. Procedures performed in the first period are repeated in the second period. Blood samples are collected pre-dose and after dosing for both treatment periods.

SECONDARY OUTCOMES:
Secondary includes the pharmokinetic parameter to measure the etanercept (ENBREL®) AUC (0-x), area under the curve | 28 days: timepoint at which outcome measure is assessed following each treatment arm
  28 days after receiving treatment in Period 1, subjects return to facility to receive the alternate treatment in Period 2. Procedures performed in the first period are repeated in the second period. (Blood samples are collected pre-dose and after dosing for both treatment periods.)
Safety Events measured by number of adverse events and retationship to treatment | 28 days following each treatment arm (total of 77 days including screening)
  Number of adverse events for each subject summarized by system organ class, severity, and relationship to treatment
Any significant changes from baseline in Vital Signs and physical examinations | Baseline and 28 days following each treatment arm (total of 77 days including screening)
  Change from baselline of vital signs, which includes blood pressure (systolic and diastolic) and heart rate per minute.
Any Clinically Significant changes in clinical laboratory tests will be noted. | Collected screening, Day -1 in both treatment periods, and day 15 in treatment period 2
  Clinically significant abnormalities in clinical laboratory tests (chemistry and hematology and urine) analyzed by standard procedures
12-lead Electrocardiograms will be performed and saved with subject source records | Performed at screening and day 15 in Treatment B
  Standard 12-lead electrocardiogram (ECG) with review of ventricular rate, rhythm, and interval measurements and appearance of the ECG waves will be performed
Blood samples obtained to measure seroreactivitiy to etanercept at baseline and following treatment | Predose in each treatment period and 28 days following dosing in treatment period B
  Blood samples to measure seroreactivity to etanercept
Secondary includes measure of pharmacokinetic parameter of Tmax, the time to reach maximum concentration | 28 days following each treatment period the outcome will be measured
  Subjects return to the facility 28 days following each treatment segment (blood samples are collected immediately pre-dose and after dosing)
Secondary outcome to measure t 1/2: elimination half-life for etanercept | Outcome to be measured 28 days following each treatment
  Subjects return to the facility 28 days following dosing; blood samples are taken immediately pre-dose and after treatment
Secondary to include etanercept pharmacokinetic parameter of CL/F: apparent clearance | Measurement assessed at 29 day timepoint following each treatment arm
  Subjects return to facility 28 days following each treatment; blood sample is obtained immediately pre-dose and after dosing

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com